CLINICAL TRIAL: NCT05703880
Title: Finerenone FIRST (Finerenone Research of Early Safety and Effectiveness), Part 2.0
Brief Title: An Observational Study Called FIRST-2.0 to Learn More About the Use of the Study Treatment Finerenone Including How Safe it is and How Well it Works Under Real-world Conditions
Acronym: FIRST-2
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 22381
Record Dates: First submitted 2023-01-20; First posted 2023-01-30 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Chronic Kidney Disease; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2 | interventions — finerenone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Finerenone (Kerendia, BAY948862): Adults with CKD and T2D from the USA who initiate finerenone.
  Interventions: Drug: Finerenone (Kerendia, BAY948862)

INTERVENTIONS:
Drug: Finerenone (Kerendia, BAY948862) — Retrospective cohort analysis using United States Optum EHR data and OM1 RWDC databases.

SUMMARY:
This is an observational study, in which data from people in the United States (US) with chronic kidney disease (CKD) together with type 2 diabetes (T2D) are studied. The participants in this study are already receiving the study treatment finerenone as part of their regular care from their doctors.

In observational studies, only observations are made without specified advice or interventions.

CKD is a long-term progressive decrease in the kidneys' ability to work properly. In people with T2D, the body does not make enough of a hormone called insulin, or does not use insulin well enough. The resulting high blood sugar levels can cause damage to the kidneys. CKD often occurs together with T2D or as a consequence of T2D.

Finerenone works by blocking certain proteins, called mineralocorticoid receptors. By doing this, it may reduce damage to kidneys, heart and blood vessels. Finerenone was recently approved in the US and is now available for doctors to prescribe to people with CKD together with T2D. Consequently, there is a need to collect more information about how finerenone is used, its safety and how well it works under real-world conditions.

The main purpose of this study is to collect and describe the characteristics of people with CKD and T2D who are receiving finerenone treatment as prescribed by their doctors. To do this, the researchers will collect data on:

* general information of the participants such as age or gender
* any other disease or medical condition in the participants
* other medications used while taking finerenone.

The researchers will also collect data on kidney function and possible heart problems to find out how well finerenone works. Additionally, medical problems possibly related to finerenone treatment will be collected to learn more about how safe finerenone is in real-world use.

The data will come from US databases Optum Electronic Health Records (EHR) and OM1 Real-World Data Cloud (RWDC). They will cover the period from July 2021 to May 2023.

Only already available data is collected and studied. There are no required visits or tests in this study.

ELIGIBILITY:
Inclusion Criteria:

* Minimum of 12 months continuous enrolment in the EHR databases with medical and pharmacy coverage measured as continuously receiving medical care from health providers contributing to the EHR system.
* No recorded prescription of finerenone prior to the index date.
* Age 18 years or older as of the index date.
* T2D diagnosis at any point before (and including) the index date using the same algorithms applicable to the specific data source as in previous studies of the FIRST program.
* CKD stages 2-4 related to eligibility will be defined according to the presence of the following criteria at any point before (and including) the index date:

  * A diagnosis code indicating CKD stage 2, 3, 4, or stage unspecified OR
  * Two Urinary Albumin-to-Creatinine Ratio (ACR) test results ≥ 30 mg/g separated by at least 90 days and no more than 540 days OR
  * Two different eGFR test results ≥ 15 mL/min/1.73 m*2 AND < 60 mL/min/1.73 m*2 separated by at least 90 days and no more than 540 days.

Exclusion Criteria:

* Type 1 diabetes identified by appropriate algorithms in the data source
* Kidney cancer on or before the index date
* Kidney failure defined as:

  * Two different eGFR test results < 15 mL/min/1.73 m*2 separated by at least 90 days and no more than 540 days
  * Dependence on dialysis (at least 3 sessions over at least 90 days during the baseline period)
  * A diagnosis code indicating kidney failure or CKD stage 5 (International Classification of Diseases, 10th Revision)
  * Kidney transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons initiating finerenone who have CKD and T2D will be included based on combinations of diagnosis codes of CKD and T2D, respectively, prescriptions and laboratory values (e.g., eGFR values or UACR measurements) indicating CKD and T2D.
Sampling Method: Non-Probability Sample
Enrollment: 15948 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Descriptive summary of characteristics of patients who initiate finerenone and have CKD and T2D in the US. | Up to 365 days
Descriptive summary of comorbidities of patients who initiate finerenone and have CKD and T2D in the US. | Up to 365 days
Descriptive summary of comedications of patients who initiate finerenone and have CKD and T2D in the US. | Up to 180 days

SECONDARY OUTCOMES:
Incidence rate of composite renal outcomes | Up to 18 months
Incidence rate of composite cardiovascular outcomes | Up to 18 months
Number of patients who initiate finerenone using a 10 mg dose and number of patients who have up-titrated to a 20 mg dose by 1, 3, 6, and 12 months, respectively. | Up to 18 months
Number of patients who initiate finerenone using a 20 mg dose and number of patients who have down-titrated to a 10 mg dose by 1, 3, 6, and 12 months, respectively | Up to 18 months
Incidence rate of hyperkalemia | Up to 18 months
Incidence of hospitalization associated with a hyperkalemia event | Up to 18 months
Change in UACR between baseline, at 4 months and end of follow up visit after initiating finerenone | Up to 18 months
  UACR: Urine Albumin to Creatinine Ratio
Change in eGFR between baseline, at 4 months and end of follow up visit after initiating finerenone | Up to 18 months
  eGFR: Estimated Glomerular Filtration Rate
Change in level of serum potassium between baseline and end of follow up visit after initiating finerenone | Up to 18 months
Incidence rates of the respective component outcomes of the CV and renal composite outcomes | Up to 18 months
Incidence rate of proliferative diabetic retinopathy in patients who initiate finerenone with prior non-proliferative diabetic retinopathy | Up to 18 months
  Proliferative diabetic retinopathy is identified by the occurrence of an inpatient or outpatient diagnosis code for proliferative diabetic retinopathy.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - OM1 Real-World Data Cloud (RWDC), Boston, Massachusetts
  - Optum electronic health records (EHR) database, Eden Prairie, Minnesota

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Derived] Vizcaya D, Kovesdy CP, Reyes A, Pessina E, Pujol P, James G, Oberprieler NG. Characteristics of patients with chronic kidney disease and Type 2 diabetes initiating finerenone in the USA: a multi-database, cross-sectional study. J Comp Eff Res. 2023 Aug;12(8):e230076. doi: 10.57264/cer-2023-0076. Epub 2023 Jun 30. PMID 37387399